CLINICAL TRIAL: NCT03565211
Title: A Prospective, Multi-Center, Non-Comparative Trial of the Clinical Safety of the Progesterone Vaginal Ring in Women Undergoing Assisted Reproductive Technology (ART) Procedures
Brief Title: Clinical Safety Study of the Progesterone Vaginal Ring in Women Undergoing Assisted Reproductive Technology Procedures
Acronym: SARA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000293
Record Dates: First submitted 2018-05-18; First posted 2018-06-21 (Actual); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-07

CONDITIONS: Progesterone Supplementation in Women Undergoing ART
Keywords: Progesterone vaginal ring (PVR); Vaginal progesterone ring; Assisted reproductive technology (ART); Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Masking Description: Open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Progesterone vaginal ring (PVR) (Experimental): Treatment started on the day following oocyte retrieval and could be continued through Week 12 of pregnancy (10 weeks post-oocyte retrieval), depending on the participants pregnancy assessment. A new PVR was inserted every 7 days with up to 10 PVRs used.
  Interventions: Drug: Progesterone vaginal ring

INTERVENTIONS:
Drug: Progesterone vaginal ring — A flexible, non-degradable PVR containing progesterone in micronized formulation and dispersed evenly throughout the ring.

SUMMARY:
The purpose of the study is to assess the safety of Progesterone Vaginal Ring (PVR) in women undergoing fresh embryo transfer (ART).

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women aged 18-34 at the time of consent.
* Documentation of a normal uterine cavity by hysteroscopy, hydrosonogram, or hysterosalpingogram within one year of screening.
* Normal Pap smear test within 24 months of screening.
* At least one cycle without reproductive hormone medication prior to screening follicle-stimulating hormone (FSH) and estradiol blood draw.
* Tubal, idiopathic, male factor, ovulatory dysfunction, or endometriosis-linked infertility.

Exclusion Criteria:

* Body mass index greater than 38 kg/m^2.
* FSH greater than 15 IU/L during the early follicular phase (Day 2-4). For those participants with polycystic ovarian syndrome, a Day 2-4 FSH level can be obtained following a progestogen withdrawal or spontaneous menses.
* Clinically significant gynecologic pathology, such as submucosal fibroids, intramural fibroids >5 cm, communicating hydrosalpinx, uncorrected uterine septum, endometrial cancer or endometrial atypia, scar tissue inside the cavity or poorly developed uterine lining from prior uterine surgery, pelvic tuberculosis, or any other conditions that could adversely affect pregnancy success.
* Uncontrolled elevation of prolactin or too little thyroid hormone in the blood.
* History of more than one failed fresh in vitro fertilization cycle. A failed cycle is defined as having started a cycle and not becoming pregnant or pregnancy loss prior to the 20th week of pregnancy.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pre-menopausal females aged 18-34 years.
Enrollment: 352 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (15):
- United States (15):
  - Fertility Treatment Center, Tempe, Arizona
  - HRC Fertility, Encino, California
  - Reproductive Associates of DE, Newark, Delaware
  - Women's Medical Research Group, Clearwater, Florida
  - Center for Reproductive Medicine, Winter Park, Florida
  - Idaho Center for Reproductive Medicine, Boise, Idaho
  - InVia Fertility, Hoffman Estates, Illinois
  - Carolina Conceptions, Raleigh, North Carolina
  - Abington Reproductive Medicine, Abington, Pennsylvania
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Center for Assisted Reproduction, Bedford, Texas
  - Houston Fertility Institute, Houston, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Utah Fertility Center, Pleasant Grove, Utah
  - Eastern Virginia Medical School | EVMS Obstetrics & Gynecology, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 14 trial centers in the United States (US) between 26 July 2018 to 29 July 2019.
Pre-assignment Details: In total 352 participants were screened. Of these, 98 were screening failures and 254 participants were treated with investigational medicinal product (IMP), progesterone vaginal ring (PVR).
Groups:
- Progesterone Vaginal Ring: Treatment started on the day following oocyte retrieval and could be continued through Week 12 of pregnancy (10 weeks post-oocyte retrieval), depending on the participants pregnancy assessment. A new PVR was inserted every 7 days with up to 10 PVRs used.
Period: Overall Study
Arm/Group | Progesterone Vaginal Ring
Started | 254
Modified Intention-to-treat (mITT) | 243 (Had successful oocyte retrieval, received >=1 dose of IMP, and completed fresh embryo transfer)
Completed | 206
Not Completed | 48
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 44
Not completed — Personal issues | 1

BASELINE CHARACTERISTICS:
Population: The safety population comprised of all participants treated with IMP.
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (2.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 224
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 17
  White | 210
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Rate of Spontaneous Abortions Occurring on or Before 12 Weeks Post-oocyte Retrieval
Description: Frequency of participants with spontaneous abortions on or before 12 weeks post-oocyte retrieval and undergoing fresh embryo transfer was presented.
  Spontaneous abortion was defined as two positive beta-human chorionic gonadotropin (β-hCG) tests occurring at least two days apart on or after 2 weeks post-oocyte retrieval, but followed by observation of any empty intrauterine gestational sac (blighted ovum), intrauterine gestation without a fetal heart beat, or absence of viable fetuses, as documented by transvaginal ultrasound (TVUS).
Time Frame: On or before 12 weeks post-oocyte retrieval
Population: The mITT analysis set consisted of all participants who had successful oocyte retrieval, received at least 1 dose of IMP, and had completed fresh embryo transfer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants | 7.4 [4.4 to 11.5]

2. Secondary Outcome: Cumulative Rate of Spontaneous Abortions Occurring at 6 Weeks Post-oocyte Retrieval
Description: Frequency of participants with spontaneous abortions at 6 weeks post-oocyte retrieval was presented.
Time Frame: At 6 weeks post-oocyte retrieval
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants | 5.8 [3.2 to 9.5]

3. Secondary Outcome: Cumulative Rate of Spontaneous Abortions Occurring at 10 Weeks Post-oocyte Retrieval
Description: Frequency of participants with spontaneous abortions at 10 weeks post-oocyte retrieval was presented.
Time Frame: At 10 weeks post-oocyte retrieval
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants | 7.4 [4.4 to 11.5]

4. Secondary Outcome: Cumulative Rate of Biochemical Abortion Within 6 Weeks Post-oocyte Retrieval
Description: Frequency of participants with biochemical abortions within 6 weeks post-oocyte retrieval was presented.
  Biochemical abortion was defined as a positive β-hCG test at 2 weeks and 2 weeks +3-4 days post-oocyte retrieval, but followed by no observed gestational sac on a later TVUS, or followed by a negative β-hCG test.
Time Frame: Within 6 weeks post-oocyte retrieval
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants | 10.3 [6.8 to 14.8]

5. Secondary Outcome: Cumulative Rate of Biochemical Abortion Within 10 Weeks Post-oocyte Retrieval
Description: Frequency of participants with biochemical abortions within 10 weeks post-oocyte retrieval was presented.
Time Frame: Within 10 weeks post-oocyte retrieval
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants | 10.3 [6.8 to 14.8]

6. Secondary Outcome: Positive β-hCG Rate at 2 Weeks and 2 Weeks +3-4 Days Post Oocyte Retrieval
Description: Frequency of participants with positive β-hCG rate at 2 weeks and 2 weeks +3-4 Days was presented. Positive β-hCG was defined as a positive serum β-hCG test at 2 weeks and 2 weeks +3-4 Days post-oocyte retrieval.
Time Frame: At 2 weeks and 2 weeks +3-4 Days post oocyte retrieval
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants | 60.9 [54.5 to 67.1]

7. Secondary Outcome: Clinical Pregnancy Rate at 6 Weeks
Description: Frequency of participants with clinical pregnancy at 6 weeks was presented. Clinical pregnancy was defined as a TVUS showing at least 1 intrauterine gestational sac with fetal heart-beat at 6 weeks post-oocyte retrieval.
Time Frame: At 6 weeks post-oocyte retrieval
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants | 44.9 [38.5 to 51.3]

8. Secondary Outcome: Clinical Pregnancy Rate at 10 Weeks
Description: Frequency of participants with clinical pregnancy at 10 weeks was presented.
Time Frame: At 10 weeks post-oocyte retrieval
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants | 43.2 [36.9 to 49.7]

9. Secondary Outcome: Rate of Ectopic and Heterotopic Pregnancies Following Oocyte Retrieval
Description: Frequency of participants with ectopic and heterotopic pregnancies was presented.
Time Frame: At 4 weeks +3-4 Days after oocyte retrieval
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 243
percentage of participants
  Ectopic pregnancy | 0.4 [0.0 to 2.3]
  Heterotopic pregnancy | 0.0 [0.0 to 1.5]

10. Secondary Outcome: Rate of Abnormal Findings in Clinical Laboratory Tests (Clinical Chemistry, Hematology, and Urinalysis)
Description: Participants with at least one abnormal finding in clinical laboratory tests (i.e. abnormal clinical significant [CS] values: as assessed by investigator) were reported. Clinical chemistry included: glucose, aspartate aminotransferase, alanine aminotransferase, blood urea nitrogen, creatinine, potassium, sodium, chloride, calcium, estimated glomerular filtration rate, and gamma-glutamyl transferase; hematology included: basophils, eosinophils, hematocrit, hemoglobin, lymphocytes, monocytes, neutrophils, platelets, erythrocytes, and leukocytes; urinalysis included: specific gravity, ketones, pH, protein, blood, and glucose.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Potassium (mmol/L)<3.5->5.3 | 1
  Blood, traces: number analyzed (Participants) | 252
  Blood, traces | 1

11. Secondary Outcome: Rate of Abnormal Findings in Vital Signs
Description: Participants with at least one abnormal finding (i.e. abnormal CS values: as assessed by investigator) in vital signs were reported. Vital signs includes: Weight (kg): decrease of >=7% from baseline (BL) or increase of >=7% from BL; Systolic Blood Pressure (SBP): <=90 mmHg and decrease of >=20 mmHg from BL or >=180 mmHg and increase of >= 20 mmHg from BL; Diastolic Blood Pressure (DBP): <= 50 mmHg and decrease of >= 15 mmHg from BL or >=105 mmHg and increase of >=15 mmHg from BL; Heart Rate: <=50 (beats per minute [bpm]) and decrease of >= 15 bpm from BL or >=120 bpm and increase of >=15 from BL; Temperature >= 38.3 degree Celsius.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Weight (kg), decrease of >=7% from BL: number analyzed (Participants) | 253
  Weight (kg), decrease of >=7% from BL | 4
  Weight (kg), increase of >=7% from BL: number analyzed (Participants) | 253
  Weight (kg), increase of >=7% from BL | 23
  SBP (mmHg), <=90 and decrease >=20 from BL | 2
  DBP (mmHg), <=50 and decrease of>=15 from BL | 3
  DBP(mmHg),>=105 and increase of>=15 from BL | 1
  Heart Rate(bpm) <=50 and decrease of>= 15 from BL | 1
  Heart Rate(bpm) >=120 and increase of>= 15 from BL | 1

12. Secondary Outcome: Frequency, Intensity/Grade, Seriousness, and Relatedness of Adverse Events (AEs)
Description: The frequency of participants with total AEs, AEs by categories of intensity (mild, moderate, severe), seriousness and relatedness was presented. An AE is any untoward medical occurrence in a participant participating in a clinical trial. The intensity of an AE was classified using the following 3-point scale: mild=awareness of signs or symptoms, but no disruption of usual activity; moderate=event sufficient to affect usual activity (disturbing); or severe= inability to work or perform usual activities (unacceptable). Seriousness refers to death, hospitalization/ prolongation of existing hospitalization, a life-threatening experience, persistent or significant disability/incapacity, or congenital anomaly. The possibility of whether the IMP caused the AE would be classified as: reasonable possibility, no reasonable possibility. All the reasonable possible causality to the IMP were referred to as adverse drug reactions (ADRs). Relatedness of AEs to IMP was assessed by the investigator.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Any AE | 124
  Mild AE | 100
  Moderate AE | 46
  Severe AE | 9
  Serious AE | 4
  ADRs | 25

13. Secondary Outcome: Frequency and Intensity/Grade of Vaginal Bleeding/Spotting
Description: Frequency of participants with vaginal bleeding/spotting was presented in total and by categories of intensity/grade (mild, moderate and severe). Vaginal bleeding was recorded in a bleeding log by the participant. The severity of the bleeding was determined using a Pictorial Blood Loss Assessment chart.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Any vaginal bleeding | 4
  Mild vaginal bleeding | 3
  Moderate vaginal bleeding | 1
  Severe vaginal bleeding | 1

14. Secondary Outcome: Frequency and Intensity/Grade of Vaginal Hemorrhage
Description: Frequency of participants with vaginal hemorrhage was presented in total and by categories of intensity/grade (mild, moderate and severe). Vaginal hemorrhage was defined as a) blood loss of greater than 500 mL based on the opinion of the Investigator or b) hemoglobin post-treatment lesser than 10 gm/dL or c) blood loss requiring transfusion.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants | 0

15. Secondary Outcome: Frequency and Intensity/Grade of Vaginal Pain
Description: The frequency of participants with vaginal pain was presented in total and by categories of intensity/grade.
  The intensity of vaginal pain was evaluated as symptoms score of pain and dyspareunia (pain with sexual activity) as: Grade 1 (mild) - Pain causing no or minimal inference with usual social & functional activities; Grade 2 (moderate) - Pain causing greater than minimal inference with usual social & functional activities or the need for non-narcotic medication; Grade 3 (severe) - Pain causing inability to perform usual social & functional activities or the need for narcotic medication; Grade 4 (potentially life threatening) - Disabling pain causing inability to perform basic self-care functions OR hospitalization (other than emergency room visit) indicated.
  Dyspareunia (pain with sexual activity): Grade 1 (mild) - Pain causing no or minimal inference with sexual function; Grade 2 (moderate) - Pain causing greater than minimal inference with sexual function.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Any vaginal pain | 2
  Mild vaginal pain | 2
  Moderate vaginal pain | 1
  Severe vaginal pain | 0
  Potentially life threatening vaginal pain | 0
  Any dyspareunia | 1
  Mild dyspareunia | 0
  Moderate dyspareunia | 1

16. Secondary Outcome: Frequency and Intensity/Grade of Vaginal Infection
Description: Frequency of participants with vaginal infection was presented in total and by categories of intensity/grade (mild, moderate and severe).
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Any vaginal infection | 4
  Mild vaginal infection | 3
  Moderate vaginal infection | 1
  Severe vaginal infection | 0

17. Secondary Outcome: Frequency and Intensity/Grade of Vaginal Irritation
Description: The frequency of participants with vaginal irritation was presented in total and by categories of intensity/grade. The intensity of vaginal irritation evaluated as symptoms score of vaginal itching, vaginal dryness, and vaginal discharge. Vaginal itching: Grade 1 (mild)-itching causing no, mild or moderate inference with usual social & functional activities; Grade 2 (moderate)-itching causing inability to perform usual social & functional activities; may require intervention such as antihistamine or bathing. Vaginal dryness: Grade 1 (mild)-dryness causing no or minimal inference with usual sexual, social & functional activities; Grade 2 (moderate)-dryness causing greater than minimal inference with usual sexual, social & functional activities. Vaginal discharge by participant report: Grade 1 (mild)-mild-moderate increase in amount above participant BL-no sanitary protection required; Grade 2 (moderate)-profuse increase in discharge requiring pad use or other hygienic intervention.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Any vaginal itching: number analyzed (Participants) | 253
  Any vaginal itching | 2
  Mild vaginal itching: number analyzed (Participants) | 253
  Mild vaginal itching | 2
  Moderate vaginal itching: number analyzed (Participants) | 253
  Moderate vaginal itching | 0
  Any vaginal dryness: number analyzed (Participants) | 252
  Any vaginal dryness | 1
  Mild vaginal dryness: number analyzed (Participants) | 252
  Mild vaginal dryness | 0
  Moderate vaginal dryness: number analyzed (Participants) | 252
  Moderate vaginal dryness | 1
  Any vaginal discharge: number analyzed (Participants) | 250
  Any vaginal discharge | 3
  Mild vaginal discharge: number analyzed (Participants) | 250
  Mild vaginal discharge | 3
  Moderate vaginal discharge: number analyzed (Participants) | 250
  Moderate vaginal discharge | 0

18. Secondary Outcome: Frequency, Intensity/Grade, Seriousness, and Relatedness of AEs Associated With Vaginal and Cervical Abrasions and Lesions
Description: Frequency of participants with AEs associated with vaginal and cervical abrasions and lesions, by intensity, seriousness, & relatedness was presented. Intensity was evaluated as symptoms score: Vaginal/cervical lesions:Grade 0 (Normal)- Normal variants including skin tags, moles, scars, etc; Grade 1 (mild) - Blisters, ulcerations, or pustules, no treatment indicated; Grade 2 (moderate)- Blisters, ulcerations, or pustules with treatment indicated; Grade 3 (severe) - Severe epithelial disruption requiring hospitalization; Vaginal/cervical abrasions: Grade 0 (Normal) - None; Grade 1 (mild)- Superficial disruptions and disruptions extending through the mucosa with minimal impact on life; Grade 2 (moderate)- Large disruptions extending through the mucosa or large superficial disruptions, hospitalization not indicated; Grade 3 (severe)- Large disruptions extending through the mucosa or large superficial disruptions, hospitalization indicated. Relatedness to IMP was assessed by investigator.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Any Vaginal lesions: number analyzed (Participants) | 253
  Any Vaginal lesions | 1
  Mild vaginal lesion: number analyzed (Participants) | 253
  Mild vaginal lesion | 1
  Moderate vaginal lesion: number analyzed (Participants) | 253
  Moderate vaginal lesion | 0
  Severe vaginal lesion: number analyzed (Participants) | 253
  Severe vaginal lesion | 0
  Serious vaginal lesion | 0
  Related vaginal lesion | 0
  Any vaginal abrasion: number analyzed (Participants) | 253
  Any vaginal abrasion | 0
  Any cervical lesion: number analyzed (Participants) | 252
  Any cervical lesion | 0

19. Secondary Outcome: Frequency, Intensity/Grade, Seriousness, and Relatedness of AEs Associated With Vaginal Adhesions
Description: The frequency of participants with AEs associated with vaginal adhesion (total), by categories of intensity, seriousness, and relatedness was presented.
  The intensity was evaluated as symptoms score of vaginal adhesion as: Grade 0 (Normal) - None; Grade 1 (mild) - asymptomatic, manual removal of ring possible; Grade 2 (moderate) - Symptomatic (eg: irritation reported by participant), manual removal of ring possible; Grade 3 (severe) - Surgical intervention (eg: adhesiolysis) required to resolve; Grade 4 (potentially life threatening) - urgent intervention indicated. The AEs associated with vaginal adhesion of Grade 4 intensity were considered to be serious. Relatedness to IMP was assessed by investigator.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 253
Participants | 0

20. Secondary Outcome: Frequency and Reason for PVR Discontinuation
Description: Frequency of participants who prematurely discontinued PVR (i.e. did not fulfill 10 weeks of PVR treatment) was presented by reason.
Time Frame: From Day 1 of PVR treatment (day after oocyte retrieval) up to end-of-trial (12 weeks post-oocyte retrieval)
Population: The safety analysis set comprised of all participants treated with IMP.
Measure: Number; unit: participants
Arm/Group | Progesterone Vaginal Ring
Number analyzed (Participants) | 254
participants
  Withdrawal by participant | 2
  Lost to follow-up | 1
  Adverse event | 44
  Personal issue | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of obtaining informed consent until the last visit (end of trial) (up to approximately 4.5 months) .
Description: Adverse events with onset after the start of the IMP administration were considered treatment-emergent and are presented for the safety analysis set.
Arm/Group | Progesterone Vaginal Ring
All-Cause Mortality (participants affected / at risk) | 0/254
Serious Adverse Events (participants affected / at risk) | 4/254
Other Adverse Events (participants affected / at risk) | 72/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone Vaginal Ring (N=254)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone Vaginal Ring (N=254)
Nausea (Gastrointestinal disorders) | 22 (22)
Headache (Nervous system disorders) | 13 (17)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 25 (25)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT03565211/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT03565211/SAP_001.pdf